CLINICAL TRIAL: NCT07275216
Title: Phase 2 Study of Pembrolizumab With Chemotherapy in Frail Patients With Newly Diagnosed Classical Hodgkin Lymphoma
Brief Title: Pembrolizumab in Combination With Chemotherapy for the Treatment of Frail Hodgkin Lymphoma Patients Ineligible for Standard Treatment
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24081; NCI-2025-08524 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24081 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Classic Hodgkin Lymphoma
MeSH Terms: interventions — Specimen Handling; Brentuximab Vedotin; Dacarbazine; Gemcitabine; pembrolizumab; Exercise Test; Magnetic Resonance Spectroscopy; Respiratory Physiological Phenomena

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (P-G, P-BV-D) (Experimental): See Detailed Description.
  Interventions: Procedure: Biospecimen Collection; Drug: Brentuximab Vedotin; Procedure: Computed Tomography; Drug: Dacarbazine; Procedure: Echocardiography Test; Drug: Gemcitabine; Biological: Pembrolizumab; Other: Physical Performance Testing; Procedure: Positron Emission Tomography; Procedure: Pulmonary Function Test

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Brentuximab Vedotin — Given IV
  Other Names: ADC SGN-35; Adcetris; Anti-CD30 Antibody-Drug Conjugate SGN-35; Anti-CD30 Monoclonal Antibody-MMAE SGN-35; Anti-CD30 Monoclonal Antibody-Monomethylauristatin E SGN-35; cAC10-vcMMAE; SGN 35; SGN-35; SGN35
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Dacarbazine — Given IV
  Other Names: 4-(Dimethyltriazeno)imidazole-5-carboxamide; 5-(Dimethyltriazeno)imidazole-4-carboxamide; Asercit; Biocarbazine; Dacarbazina; Dacarbazina Almirall; Dacarbazine - DTIC; Dacatic; Dakarbazin; Deticene; Detimedac; DIC; Dimethyl (triazeno) imidazolecarboxamide; Dimethyl Triazeno Imidazol Carboxamide; Dimethyl Triazeno Imidazole Carboxamide; dimethyl-triazeno-imidazole carboxamide; Dimethyl-triazeno-imidazole-carboximide; DTIC; DTIC-Dome; Fauldetic; Imidazole Carboxamide; Imidazole Carboxamide Dimethyltriazeno; WR-139007
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
Other: Physical Performance Testing — Ancillary studies
  Other Names: Physical Fitness Testing; Physical Function Testing
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Procedure: Pulmonary Function Test — Ancillary studies
  Other Names: lung function test; PFT; Pulmonary Function Testing; Pulmonary Function Tests

SUMMARY:
This phase II trial tests how well pembrolizumab in addition to chemotherapy (gemcitabine, brentuximab vedotin, and dacarbazine) works in treating frail patients with newly diagnosed Hodgkin lymphoma who aren't candidates for standard anthracycline-based treatment. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of cancer cells to grow and spread. Gemcitabine is a chemotherapy drug that blocks the cells from making deoxyribonucleic acid (DNA) and may kill cancer cells. Brentuximab vedotin is in a class of medications called antibody-drug conjugates. It is made of a monoclonal antibody called brentuximab that is linked to a cytotoxic agent called vedotin. Brentuximab attaches to CD30 positive lymphoma cells in a targeted way and delivers vedotin to kill them. Dacarbazine is in a class of medications called alkylating agents. It works by damaging the cell's DNA and may kill cancer cells and slow down or stop cancer growth. Pembrolizumab in combination chemotherapy may be a safe and effective alternative treatment option for frail patients with Hodgkin lymphoma who can't receive standard anthracycline-based treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Estimate the best complete metabolic response (CMR) rate for frail patients with classical Hodgkin lymphoma (cHL) who receive pembrolizumab and gemcitabine (P-G).

SECONDARY OBJECTIVES:

I. Estimate CMR rate, overall response rate (ORR), progression-free-survival (PFS), duration of response (DOR), and overall response (OS) among patients who receive P-G (± pembrolizumab maintenance).

II. Estimate CMR, overall response, PFS, DOR, and OS among patients who receive pembrolizumab, brentuximab vedotin, and dacarbazine (P-BV-D).

III. Evaluate the toxicity of P-G, pembrolizumab maintenance, and P-BV-D.

EXPLORATORY OBJECTIVES:

I. Explore association between geriatric assessment measures (Cancer and Aging Research Group [CARG] geriatric assessment) and toxicity and efficacy in the elderly patients enrolled on this trial.

II. Assess functional trajectory determined by short physical performance battery (SPPB) change score in the elderly patients enrolled on this trial.

III. Explore the association between clinical outcomes and pathological tumor characteristics.

OUTLINE:

CYCLES 1-8: Patients receive pembrolizumab intravenously (IV) over 30 minutes and gemcitabine IV on day 1 of each cycle. Cycles repeat every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. Patients without progressive disease during or at the completion of 8 cycles of P-G proceed to maintenance therapy. Patients with progressive disease during or at the completion of 8 cycles of P-G proceed to salvage therapy.

MAINTENANCE THERAPY: Patients receive pembrolizumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 42 days for up to 4 cycles (cycles 9-12) in the absence of disease progression or unacceptable toxicity.

SALVAGE THERAPY: Patients receive pembrolizumab IV over 30 minutes, brentuximab vedotin IV over 30 minutes, and dacarbazine IV on day 1 of each cycle. Cycles repeat every 21 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

Patients undergo positron emission tomography (PET)/computed tomography (CT) and collection of blood samples throughout the trial and may undergo echocardiography (ECHO) at screening if indicated.

After completion of study treatment, patients are followed up at 30 days and at 12, 18 (salvage patients), and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Meets at least one of the following criteria indicating unsuitability for conventional anthracycline-based frontline chemotherapy, as determined by the investigator:

  * Age ≥ 75 years
  * Eastern Cooperative Oncology Group (ECOG) 2-4
  * Left ventricular ejection fraction (LVEF) < 50%
  * Creatinine clearance < 60 mL/min, using Cockcroft-Gault formula or equivalent
  * Pulmonary function impairment: forced expiratory volume in 1 second (FEV1) < 50% and/or diffusion capacity of the lung for carbon monoxide (DLCO) < 50%
* ECOG ≤ 2
* Age ≥ 18 years
* Histologically confirmed new diagnosis of classical Hodgkin lymphoma (excluding nodular lymphocyte predominant Hodgkin lymphoma) according to the World Health Organization (WHO) classification, with hematopathology review at the participating institution
* No prior systemic treatment for classical Hodgkin lymphoma with the following exceptions: a course of systemic corticosteroids for palliation of symptoms related to the classical Hodgkin lymphoma is allowed but must be stopped by cycle 1 day 1 (C1D1) as well as prior treatment with P-G as part of this clinical trial for patients will receive P-BV-D
* Measurable disease (at least one non-bone fludeoxyglucose F-18 [FDG]-avid lesion ≥ 1.5 cm in long axis)
* Absolute neutrophil count (ANC) ≥ 1,000/mm^3

  * NOTE: Growth factor is not permitted within 7 days of ANC assessment unless cytopenia is secondary to disease involvement
* Platelets ≥ 50,000/mm^3

  * NOTE: Platelet transfusions are not permitted within 7 days of platelet assessment unless cytopenia is secondary to disease involvement
* Total bilirubin ≤ 2 × upper limit of normal (ULN) or direct bilirubin ≤ 2 × ULN for patients with Gilbert's disease
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x ULN
* AST and ALT ≤ 3 x ULN unless there is liver involvement by lymphoma in which case AST and ALT < 5 x ULN
* For patients for whom P-BV-D therapy is planned, creatinine clearance of ≥ 30 mL/min per 24-hour urine test or the Cockcroft-Gault formula
* If not receiving anticoagulants: International normalized ratio (INR) OR prothrombin (PT) ≤ 1.5 x ULN

  * If on anticoagulant therapy: PT must be within therapeutic range of intended use of anticoagulants
* If not receiving anticoagulants: Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN

  * If on anticoagulant therapy: aPTT must be within therapeutic range of intended use of anticoagulants
* Seronegative for hepatitis C virus (HCV), hepatitis B virus (HBV) (surface antigen negative) OR

  * If seropositive for HBV or HCV, nucleic acid quantitation must be performed. Viral load must be undetectable. Patients with occult or prior HBV infection (defined as negative hepatitis B virus surface antigen [HBsAg] and positive hepatitis B core antibody [HBcAb]) may be included if HBV DNA is undetectable, if they are willing to undergo DNA testing on day 1 of every cycle and every three months for at least 12 months after the last cycle of study treatment
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* A male participant must agree to use a contraception during the treatment period and for at least 6 months after the last dose of study treatment and refrain from donating sperm during this period
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) OR
  * A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least (X days/weeks [corresponding to time needed to eliminate any study treatment(s)] [pembrolizumab and/or any active comparator/combination] plus 30 days [a menstruation cycle] for study treatments with risk of genotoxicity) after the last dose of study treatment
* TO PROCEED WITH SALVAGE TREATMENT: ECOG ≤ 2
* TO PROCEED WITH SALVAGE TREATMENT: Resolution of treatment-related adverse events (AEs) to baseline or grade 1, whichever is higher
* TO PROCEED WITH SALVAGE TREATMENT: Measurable disease (at least one non-bony FDG-avid lesion ≥ 1.5 cm in long axis)
* TO PROCEED WITH SALVAGE TREATMENT: Peripheral neuropathy ≤ grade 2
* TO PROCEED WITH SALVAGE TREATMENT: ANC ≥ 1,000/mm^3

  * NOTE: Growth factors are permitted
* TO PROCEED WITH SALVAGE TREATMENT: Platelets ≥ 50,000/mm^3

  * NOTE: Platelet transfusions are permitted
* TO PROCEED WITH SALVAGE TREATMENT: Hemoglobin ≥ 8 g/dL (no transfusion allowed within 3 days prior to screening)
* TO PROCEED WITH SALVAGE TREATMENT: Total bilirubin ≤ 2 x ULN or direct bilirubin ≤ 2 x ULN for patients with Gilbert's disease
* TO PROCEED WITH SALVAGE TREATMENT: AST ≤ 3 x ULN, or less then 5 x ULN for patients with liver involvement by lymphoma
* TO PROCEED WITH SALVAGE TREATMENT: ALT ≤ 3 x ULN, or less then 5 x ULN for patients with liver involvement by lymphoma
* TO PROCEED WITH SALVAGE TREATMENT: Creatinine clearance of ≥ 30 mL/min per 24-hour urine test or the Cockcroft-Gault formula

Exclusion Criteria:

* Concomitant investigational therapy
* Live vaccine within 30 days prior to day 1 of protocol therapy (e.g. measles, mumps, rubella, varicella, yellow fever, rabies, Bacille Calmette Guerin [BCG], oral polio vaccine, and oral typhoid)
* Grade ≥ 2 peripheral neuropathy
* Requirement for hemodialysis or peritoneal dialysis. Estimated glomerular filtration rate (EGFR) > 30 for pembrolizumab + BV + dacarbazine
* Known active central nervous system (CNS) involvement by lymphoma including parenchymal and/or lymphomatous meningitis
* History of prior ≥ grade 3 hypersensitivity to either brentuximab vedotin or pembrolizumab
* Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment)
* History of another primary malignancy that has been in remission for fewer than 3 years, with the following exceptions:

  * Non-melanoma skin cancer treated with curative intent
  * In situ cervical cancer
  * If the malignancy is expected to not require any systemic treatment for at least 2 years (this exception should be discussed with the study PI)
* Condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days of study drug administration. Exceptions are:

  * Inhaled or topical steroids and
  * Adrenal replacement doses > 10 mg daily prednisone equivalents in the absence of active autoimmune disease
  * Up to 7 days of 20 mg daily prednisone equivalent after C1D1 for management of lymphoma-related symptoms
* History of progressive multifocal leukoencephalopathy (PML)
* Active pneumonitis or interstitial lung disease
* Prior solid organ or allogeneic stem cell transplantation
* History of known or suspected hemophagocytic lymphohistiocytosis (HLH)
* Active, known or suspected autoimmune disease. The following are exceptions:

  * Vitiligo
  * Psoriasis not requiring systemic treatment
  * Hemolytic anemia associated with the lymphoma
  * Type I diabetes mellitus, if adequately controlled with therapy
  * Thyroid disease, if adequately controlled with therapy
  * Conditions not expected to recur in the absence of an external trigger (such exceptions should be discussed with the study PI)
* Active history of:

  * Hepatitis B (HBV) or C (HCV) infection. Patients with past HBV infection (defined as negative HBsAg and positive hepatitis B core antibody [HBcAb]) are eligible if HBV DNA is undetectable. Patients who are positive for HCV antibody are eligible if polymerase chain reaction (PCR) is negative for HCV RNA
* HIV positive
* History of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction, or cardiac symptoms consistent with New York Heart Association class III-IV within 6 months prior to day 1 of protocol therapy
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Complete metabolic response (CMR) to pembrolizumab and gemcitabine (P-G) | During/after cycles 1-8 of P-G (cycle length = 21 days), before initiation of salvage or maintenance therapy or non-protocol lymphoma therapy
  Will be estimated by the proportion of response-evaluable patients achieving a best response of CMR, along with the 95% exact binomial confidence interval.

SECONDARY OUTCOMES:
CMR | During/after cycles 1-8 of P-G (cycle length = 21 days) or cycles 1-4 of pembrolizumab maintenance (cycle length = 42 days), before initiation of non-protocol lymphoma therapy
  Will be estimated by the proportion of response-evaluable patients achieving a best response of CMR, along with the 95% exact binomial confidence interval.
Overall response (OR) | During/after cycles 1-8 of P-G (cycle length = 21 days) or cycles 1-4 of pembrolizumab maintenance (cycle length = 42 days), before initiation of non-protocol lymphoma therapy
  Will be estimated by the proportion of response-evaluable patients achieving a best response of CMR or partial metabolic response (PMR), along with the 95% exact binomial confidence interval.
Progression-free survival (PFS) | From start of P-G treatment to time of disease relapse/progression or death, assessed up to 24 months
  Will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% confidence interval will be constructed based on log-log transformation. Median value will be estimated when available.
Duration of response (DOR) | From first achievement of CMR or PMR during/after cycles 1-8 of P-G (cycle length = 21 days) or cycles 1-4 of pembrolizumab maintenance (cycle length = 42 days) to disease relapse/progression or death, assessed up to 24 months
  Will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% confidence interval will be constructed based on log-log transformation. Median value will be estimated when available.
Overall survival (OS) | From start of P-G treatment to time of death, assessed up to 24 months
  Will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% confidence interval will be constructed based on log-log transformation. Median value will be estimated when available.
Incidence of adverse events | Up to 24 months
  Toxicities will be coded and graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Event (CTCAE) version (v) 5.0. Observed toxicities of study therapy will be summarized by type (organ affected or laboratory determination such as absolute neutrophil count), severity, and attribution.
CMR (for patients who receive salvage therapy) | During/after cycles 1-12 of pembrolizumab, brentuximab vedotin, and dacarbazine (P-BV-D) (cycle length = 21 days), before initiation of non-protocol lymphoma therapy
  Will be estimated by the proportion of response-evaluable patients achieving a best response of CMR, along with the 95% exact binomial confidence interval.
OR (for patients who receive salvage therapy) | During/after cycles 1-12 of P-BV-D (cycle length = 21 days), before initiation of non-protocol lymphoma therapy
  Will be estimated by the proportion of response-evaluable patients achieving a best response of CMR or PMR, along with the 95% exact binomial confidence interval.
PFS (for patients who receive salvage therapy) | From start of P-BV-D treatment to time of disease relapse/progression or death, assessed up to 24 months
  Will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% confidence interval will be constructed based on log-log transformation. Median value will be estimated when available.
DOR (for patients who receive salvage therapy) | From first achievement of CMR or PMR during/after cycles 1-12 of P-BV-D (cycle length = 21 days) to disease relapse/progression or death, assessed up to 24 months
  Will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% confidence interval will be constructed based on log-log transformation. Median value will be estimated when available.
OS (for patients who receive salvage therapy) | From start of P-BV-D treatment to time of death, assessed up to 24 months
  Will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% confidence interval will be constructed based on log-log transformation. Median value will be estimated when available.
Incidence of adverse events (for patients who receive salvage therapy) | Up to 24 months
  Toxicities will be coded and graded using the NCI CTCAE v 5.0. Observed toxicities of study therapy will be summarized by type (organ affected or laboratory determination such as absolute neutrophil count), severity, and attribution.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Mei, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States